CLINICAL TRIAL: NCT00467012
Title: Phase Ⅱ Clinical Study of R435 (Bevacizumab) in Combination With Paclitaxel in Patients With Inoperable Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JO19901
Record Dates: First submitted 2007-04-26; First posted 2007-04-27 (Estimated); Last update posted 2012-04-26 (Estimated); Status verified 2012-04

CONDITIONS: Metastatic Breast Cancer
Keywords: Inoperable metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- step 1 (Experimental): 6 enrollment for 1 cycle(4 weeks)
  Interventions: Drug: bevacizumab; Drug: Paclitaxel
- step 2 (Experimental): 114 enrollment through to meet the stopping criteria
  Interventions: Drug: bevacizumab; Drug: Paclitaxel

INTERVENTIONS:
Drug: bevacizumab — 10mg/kg，Day1, 15 of 1 cycle(4 weeks)
Drug: Paclitaxel — 90mg/ m2，Day1, 8, 15 of 1 cycle(4 weeks)

SUMMARY:
To investigate the efficacy, safety, and pharmacokinetics when R435 and paclitaxel are administered concomitantly to patients with metastatic breast cancer.

ELIGIBILITY:
* At least 20 years old and obtained a written informed consent
* Advanced breast cancer (StageⅣ) or Inoperable metastatic breast cancer
* HER2 negative
* At least one measurable lesion based on RECIST criteria
* No previous chemotherapy for metastatic breast cancer

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2007-04; Primary Completion 2009-06 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Safety | throughout study
Progression-free survival (PFS) | event driven

SECONDARY OUTCOMES:
Overall Survival(OS) | event driven
Time to Treatment Failure(TTF) | evnt driven
Response Rate(RR) | event driven

CONTACTS AND LOCATIONS:
Overall Officials: Shingo Koganezawa, Study Chair — Clinical research department 3
Locations (5):
- Japan (5):
  - Kanto Region, Kanto
  - Kinki Region, Kinki
  - Kyushu region, Kyushu
  - Sikoku region, Sikoku
  - Tohoku region, Tōhoku